CLINICAL TRIAL: NCT04499573
Title: Safety and Efficiency of Anti-CD19/CD22 Tandem Fully Human Chimeric Antigen Receptor (CAR)-Transduced T-cell Therapy for Pediatric and Young Adult Patients With Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia: a Single Centre, Non-randomised, Open Label Phase I-II Clinical Trial of Automatically Produced Cell Therapy Product MB-CAR-T19-22 Using CliniMACS Prodigy
Brief Title: Bispecific CD19/CD22 CAR-T for Treatment of Children and Young Adults With r/r B-ALL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCPHOI-2020-07
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: B-ALL
Keywords: B-ALL; acute lymphoblastic leukemia; CAR-T
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Cyclophosphamide; Cytarabine; Etoposide; Dexamethasone; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention/treatment (Experimental): Intervention:
  1. Patient (cohort 1 and 2) or donor (cohort 3) leukapheresis
  2. Drug therapy:
     * Fludarabine 120 mg/m2
     * Cyclophosphamide 750 mg/m2
     * Etoposide 450 mg/m2
     * Cytarabine 900 mg/m2
     * Dexamethasone 30 mg/m2
     * Tocilizumab 8 mg/kg BW
  3. Biological:
  Cohort 1 and 2: autologous CD19/CD22 CAR-T lymphocytes, dose 0.15 - 1.5х106/kg
  Cohort 3: allogeneic CD19/CD22 CAR-T lymphocytes, dose 0.1х106/kg + allogeneic HSCT from a haploidentical or matched related donor
  Interventions: Drug: CD19/CD22 CAR-T

INTERVENTIONS:
Drug: CD19/CD22 CAR-T — The treatment plan will be based on stratification by the initial leukemia burden.
  Patients with "low disease burden" will receive a lymphodepletion chemotherapy of fludarabine (total dose 120mg/m2) and cyclophosphamide (total dose 750mg/m2) over 5 days.
  Patients will "high disease burden" will receive a lymphodepletion chemotherapy of fludarabine (total dose 120 mg/m2), cyclophosphamide (total dose 750 mg/m2), cytarabine (total dose 900 mg/m2), etoposide (total dose 450 mg/m2), dexamethasone (total dose 30 mg/m2) over 5 days.
  Based on interim analysis the following dosing approach will be implemented starting April 2021:
  Cohort 1: CD19+ disease, low and high burden: 1st dose - 150k/kg, 2nd dose - 850k/kg Cohort 2: CD19- disease, low and high burden: 1st dose - 500k/kg, 2nd dose - 500k/kg Cohort 3: HSCT+CAR-T: 100k/kg
  Other Names: Fludarabine; Cyclophosphamide; Cytarabine; Etoposide; Dexamethasone; Tocilizumab; Allogeneic HSCT

SUMMARY:
The purpose of this study is to evaluate the safety and efficiency of autologous CD19/CD22 CAR-T lymphocytes in a cohort of pediatric and young adult patients with relapsed /refractory B-lineage acute lymphoblastic leukemia

DETAILED DESCRIPTION:
The main objectives of the study are:

* To investigate the incidence of adverse events of grade 3-5 within after CD19/CD22 CAR lymphocyte infusion by day 28,
* To evaluate the incidence of complete remission and MRD-negative CR by day 28
* To evaluate the long-term effectiveness of CD19/CD22 CAR-T therapy (cumulative incidence of relapse, event-free survival, overall survival) at 1, 2, and 5 years after infusion.
* To evaluate the persistence of CD19/CD22 CAR-T cells and duration of B-cell aplasia (<1% B-cells in the blood) and hypogammaglobulinemia In order to prevent the development of CRS, all patients will receive an infusion of tocilizumab at 8 mg/kg body weight on day 0 before CAR-T cells infusion.

Step-down and step-up dosing will be used to adapt the trial to the scenario of excess toxicity and/or suboptimal effect. Reevaluation of dosing will be done for each cohort separately after the enrollment 5th study subject reaches day 28 or earlier if the threshold for excess toxicity or suboptimal effect is achieved.

Based on interim analysis in March 2021 after the enrollment 5th study subject reaches day 28 study population will be divided into three cohorts:

1. CD19-positive (both CD19 and CD22 expressed on over 50% of leukemia cells), low and high disease burden.
2. CD19-negative (CD22 expressed on over 50% of leukemia cells) low and high disease burden;
3. Allogeneic HSCT+ allogeneic CAR-T cohort

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent (for patients > 14 years old). For subjects < 18 years old their legal guardian must give informed consent
* CD19 or CD22 expression must be detected on greater than 50% of leukemic cells by flow cytometry
* Presence of a measurable mass of tumor cells in the bone marrow or extramedullary sites at the time of patient's inclusion in the study
* Patients with relapsed or refractory CD19 and CD22-expressing B-cell ALL:

  * Induction failure
  * MRD ≥ 0,1% after 2nd chemotherapy course for high-risk group patients.
  * First bone marrow or combined relapse of acute lymphoblastic leukemia, no CR or MRD ≥ 0,1% after 1-course 2nd line therapy
  * Second and further relapse of ALL
  * Relapse or MRD ≥ 0,1% of ALL after hematopoietic stem cell transplant (> 60 days post alloHSCT)o There must be no available alternative approved curative therapies
* Patient Clinical Performance Status: Karnofsky >50% or Lansky >50%
* Patient Life Expectancy > 4 weeks
* Patients recovered from acute toxic effects of prior chemotherapy, immune- or radiotherapy
* Patient absolute blood naïve (CD45RA+) T-lymphocyte count ≥ 50/mm3
* Patient cardiac function left ventricular ejection fraction greater than or equal to 40% by MUGA or cardiac MRI, or fractional shortening greater than or equal to 28% by ECHO or left ventricular ejection fraction greater than or equal to 50% by ECHO.
* Patients who agree to long-term follow up for up to 5 years (if received CD19/CD22 CAR-T cell infusion)
* March 2021 amendment: Healthy HLA-matched related or haploidentical donor (only for HSCT cohort)

Exclusion Criteria:

* <50% expression of both CD19 and CD22 on the leukemic population
* Active (detectable viremia) hepatitis B, C or HIV infection
* Oxygen saturation ≤ 90%
* Bilirubin >3x upper norma limit
* Creatinine >3x upper norma limit
* Active acute GVHD overall grade ≥2 (Seattle criteria)
* Moderate/severe chronic GVHD (NIH consensus) requiring systemic steroids
* Clinical signs of grade > 3 CNS disorders (seizure disorder, paresis, aphasia, cerebrovascular, ischemia/hemorrhage, severe brain injuries, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder)
* Pregnant or lactating women.
* Active (unresolved) severe infection

Ages: 3 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
incidence of grade 3-5 SAE | 1 month
  Safety:
  Toxicity evaluation following CD19/CD22 CAR T-cell infusion:
  - incidence of grade 3-5 SAE (according CTCAE v.5.0)
incidence of grade 3-5 Severe Cytokine Release Syndrome | 1 month
  Safety:
  Toxicity evaluation following CD19/CD22 CAR T-cell infusion:
  - incidence of grade 3-5 Severe Cytokine Release Syndrome (according ASTCT consensus)
incidence of grade 3-5 ICANS | 1 month
  Safety:
  Toxicity evaluation following CD19/CD22 CAR T-cell infusion:
  - incidence of grade 3-5 ICANS (according to ASTCT consensus)
Rate of complete remission | 1 month
  Efficacy:
  - Rate of complete remission among all enrolled patients (Intent-to-Treat population)
Rate of MRD-negative remission | 1 month
  Efficacy:
  - Rate of MRD-negative remission among all patients (Intent-to-treat population)
March 2021 amendment: incidence of graft failure before day 100 (only for HSCT cohort) | 100 days
  Safety:
March 2021 amendment: incidence of aGVHD grade 2-4 (only for HSCT cohort) | 100 days
  Safety:

SECONDARY OUTCOMES:
Duration of MRD-negative remission | 2 years
  Efficacy:
Persistence/frequency of CD19/CD22 lymphocytes in peripheral blood (flow cytometry) | 2 years
  Efficacy:
Duration of B-cell aplasia and hypogammaglobulinemia | 2 years
  Efficacy:
Overall survival | 5 years
  Efficacy:
Safety and adverse effects long-term | 5 years
  Safety:
March 2021 amendment: Incidence of chronic GVHD (only for HSCT cohort) | 5 years
  Safety:

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maschan, Principal Investigator — National Research Center for Pediatric Hematology , Moscow, Russian Federation
Locations (1):
- Federal Research Institute of Pediatric Hematology, Oncology and Immunology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided